CLINICAL TRIAL: NCT02842489
Title: The Role of Left Lateral Tilt-down Position During Colonoscopy Insertion: a Randomized Controlled Trial
Brief Title: Left Lateral Tilt-down Position During Colonoscopy Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept and Digestive Endoscopy Center, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: body position-1
Record Dates: First submitted 2016-06-26; First posted 2016-07-25 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Colonoscopy Insertion
Keywords: colonoscopy insertion; tilt-down position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- left lateral tilt-down position (Experimental): patients will be positioned on left lateral tilt-down position during colonoscopy until sigmoid-descending junction were examined, and then patients will be positioned on the left lateral horizontal position during colonoscopy
  Interventions: Procedure: left lateral tilt-down position
- left lateral horizontal body position (Active Comparator): patients will be positioned on the left lateral horizontal position during colonoscopy insertion
  Interventions: Procedure: left lateral horizontal position

INTERVENTIONS:
Procedure: left lateral tilt-down position — patients will be positioned on their left side and at an angle of 20 degree
  Arms: left lateral tilt-down position
Procedure: left lateral horizontal position — patients will be horizontally positioned on their left side
  Arms: left lateral horizontal body position

SUMMARY:
The purpose of this study is to determine whether the left lateral tilt-down position, which includes procedures that involve placing patients on their left lateral side at an angle to make their heads lower than their feet, is more beneficial than the left lateral horizontal body position (patient horizontally laying on their left side, traditionally used for colonoscopies) to decrease descending colon insertion time, the difficulty of colonoscopy procedure and patients' pain.

DETAILED DESCRIPTION:
Supine with tilt-down position (trendelenburg position) is used in abdominal and gynecological surgery to allow better access to the pelvic organs, as gravity pulls the bowel out of the pelvic cavity and the rectosigmoid angle straightens, which may also be favorable for colonoscopy insertion. However, few published studies have explored the value of tilt-down position in the colonoscopy (left lateral horizontal body position are usually used) and there is consequently little evidence to support left lateral tilt-down position or left lateral horizontal body position. So the investigators perform a randomized controlled trial of left lateral tilt-down position versus left lateral horizontal position for colonoscopy to investigate the safety and efficacy of lateral tilt-down position.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose age is between 18-75
2. Patients who have indications for diagnostic or therapeutic colonoscopy .
3. Patients who have signed inform consent form

Exclusion Criteria:

1. Patients who have undergone colonic resection
2. Patients with glaucoma
3. Patients with intracranial and/or central nervous system disease, including cerebral infarction and cerebral hemorrhage.
4. Patients with severe chronic cardiopulmonary and renal disease.
5. Patients with uncontrolled acid reflux disease or active nausea/vomiting.
6. Patients who are unwilling or unable to consent.
7. Patients who are not suitable for colonoscopy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
cecal colon insertion time | This outcome is measured when cecal colon is intubated during a colonoscopy

SECONDARY OUTCOMES:
patients' discomfort of colonoscopy | 2 hours
  patients' discomfort will be assessed by a 10-cm visual analog scale
endoscopists' perception of difficulty of colonoscopy | 2 hours
  difficulty of colonoscopy will be assessed by a 10-cm visual analog scale
decending insertion time | This outcome is measured when decending colon is intubated during a colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhaoshen, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

REFERENCES:
- [Derived] Zhao SB, Yang X, Fang J, Wang SL, Gu L, Xia T, Su XJ, Wang D, Li ZS, Bai Y. Effect of left lateral tilt-down position on cecal intubation time: a 2-center, pragmatic, randomized controlled trial. Gastrointest Endosc. 2018 Mar;87(3):852-861. doi: 10.1016/j.gie.2017.11.012. Epub 2017 Nov 20. PMID 29158180